CLINICAL TRIAL: NCT06145503
Title: The Effect of Dance Intervention on Cognitive Functions and Quality of Life in Patients With Chronic Stroke: A Single-Blind Randomized Controlled Study
Brief Title: Dance Intervention on Cognitive Functions and Quality of Life in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Asst. Prof., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCS20062023
Record Dates: First submitted 2023-11-16; First posted 2023-11-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Impairment; Stroke; Quality of Life
Keywords: Cognitive impairment; Dance; Stroke; Quality of life
MeSH Terms: conditions — Cognitive Dysfunction; Stroke

STUDY DESIGN:
Intervention Model Description: The sample size was determined as 36 chronic stroke patients in total (18 for each group) for the two groups (dance intervention group, control group) with an effect size of 1,000 and a targeted test power of 0.90 (90%) in the G*Power 3.1.9.6 program with an error of α=0.05 and a reference to a previous study on the subject. During the course of the research, and in anticipation of potential dropouts or patient mortality, the sample size for each group was increased, resulting in a total of 40 chronic stroke patients, with 20 patients in each group, being included in the study.
Who Masked: Participant
Masking Description: In this single-blind, randomized, controlled clinical trial, certain measures were taken to minimize bias throughout the study. The researcher responsible for collecting data from the participants with chronic stroke was unaware of the patient's allocation to either the intervention or control groups. Simultaneously, the principal investigator in charge of the dance intervention group remained blinded to the initial assessments conducted for both the dance intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance Intervention Group (Experimental): Patients within the dance intervention group (n=20) were initially required to complete a "Patient Information Form" and provide written informed consent following an explanation of the study. Over the course of 12 weeks, these patients (n=20) received a 60-minute dance intervention three times a week, led by a dance instructor. Assessments, including the "MoCA" and "SS-QOL," were conducted three times: before the dance intervention (pre-test/0th week), at the 6th week (interim measurement), and after completing the 12-week study (post-test/12th week).
  Interventions: Device: Dance Intervention Group
- Control Group (No Intervention): The control group did not receive any intervention beyond participating in data collection. Patients in this group underwent assessments with the "MoCA" and "SS-QOL" before the study (pre-test/0th week), at the 6th week of the study (interim measurement), and after the completion of the 12-week study (post-test/12th week).

INTERVENTIONS:
Device: Dance Intervention Group — The dance sessions, tailored to participants' preferences, were accompanied by music from the 80s and 90s. A dance instructor demonstrated each dance step, and the sessions comprised a 10-minute warm-up, 40 minutes of dancing, and a 10-minute cool-down. The complexity and intensity of the dance routines were adjusted based on individual abilities, functional variations, and capacity.
  Arms: Dance Intervention Group

SUMMARY:
To examine the effect of dance interventions on cognitive functions and quality of life in patients with chronic stroke.

DETAILED DESCRIPTION:
Stroke is a prevalent medical condition, primarily affecting individuals aged 65 and older. However, it can also strike young people and even children and ranks as the second leading cause of non-traumatic disability and cognitive impairment among adults. Stroke can lead to a range of physical, sensory, and cognitive deficits and impairments in psychosocial functioning. One of the most significant challenges faced by stroke survivors is cognitive impairment. The prevalence of cognitive impairment following a stroke varies widely, ranging from 20% to 80%, and it is influenced by factors such as geographical location, ethnicity, and diagnostic criteria. Stroke can disrupt various cognitive functions, including information processing, memory, planning, problem-solving, spatial awareness, apraxia, motor control, spatial perception, confusion, denial (anosognosia), and object recognition issues (agnosia). The literature reports that 30% of stroke patients experience functional limitations related to balance, speech, and cognitive issues. Particularly, more than half of stroke patients over the age of 65 experience hemiparesis, and around 30% require assistance for walking. Chronic stroke can also lead to balance and mobility problems, affecting daily life activities and significantly impacting the patient's overall quality of life.

There is a growing need for improvements in the post-stroke experience and long-term care for stroke patients. In this context, rehabilitation interventions play a vital role. Rehabilitation interventions aim to prevent complications, reduce neurological deficits, maximize functional capacity, and ultimately promote personal autonomy and social integration. Dance intervention, as part of the rehabilitation process, is recognized as an effective approach to addressing chronic stroke-related motor disorders, positively impacting post-stroke health, and promoting socialization. Dance, characterized by rhythmic body movements to music, serves as a form of artistic or emotional expression and can be performed individually, in pairs, or in groups. It is a multifaceted activity that engages both physical and cognitive abilities. Dance has been found to have positive effects on emotions, sensory stimulation, motor coordination, social interaction, perception, executive functions, and memory. Literature suggests that dance intervention helps to improve both the physical and cognitive impairments of stroke patients through promoting interpersonal harmony and multiple stimulations, and therefore its use is recommended to enhance the cognitive and physical functions of chronic stroke patients. In light of this information, this single-blind, randomized, controlled study aims to investigate the impact of dance intervention on cognitive functions and quality of life among chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria

* Being over 18 years of age,
* Volunteering to participate in the study,
* Clear consciousness and be able to communicate,
* Hemorrhagic or ischemic stroke at least 6 months ago,
* Ability to walk 10 meters without physical assistance and tolerate 50 minutes of exercise,
* Standing, maintaining balance,
* Not having had more than one stroke attack,
* A score of 21 or lower on the Montreal Cognitive Assessment Scale (MoCA).

Exclusion criteria Exclusion criteria were not meeting the inclusion criteria, having a known psychological disorder, having orthopedic disorders, having severe cognitive impairment, having an affected gait and balance, having undergone a recent surgical operation, having hearing loss, and having additional neurological diseases other than stroke.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The Montreal Cognitive Assessment | 12 Weeks
  The Montreal Cognitive Assessment (MoCA) is a cognitive assessment tool designed to evaluate cognitive functions, especially in the early stages of cognitive impairment. The MoCA scale is scored between 0 and 30 points, with higher scores indicating better cognitive functioning.
  A significant increase was found in the "MoCA" general score averages in the dance intervention group.
The Stroke Specific Quality of Life Scale | 12 Weeks
  The "Stroke Specific Quality of Life Scale (SS-QOL)" is a five-point Likert-type scale (1 point = "Strongly agree" - 5 points = "Strongly disagree"). The total score of the scale is calculated by summing the average scores from each of the 12 domains and dividing by 12. A higher total scale score signifies a higher quality of life, while a lower score indicates a lower quality of life.
  The mean scores of the dance intervention group on the activities, social and family roles, language, energy, mood, personality, thinking sub-dimensions, and total of the SS-QOL increased significantly from pre-test to post-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Tecnical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later